CLINICAL TRIAL: NCT05334966
Title: Evaluation of the Use of Supplemental Oxygen to Mothers With Fetal Left Heart Hypoplasia
Brief Title: Maternal Hyperoxygenation in Fetal Left Heart Hypoplasia
Acronym: MHO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Shaine Morris, Associate Professor, Baylor College of Medicine
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-33802
Record Dates: First submitted 2015-05-04; First posted 2022-04-19 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Left Heart Hypoplasia
MeSH Terms: interventions — Oxygen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Historical LHH Controls (No Intervention): Previous women with a dx of fetal LHH and whose care was continued at Texas Children's Hospital.
- Healthy Fetal Controls (Placebo Comparator): Healthy mothers with healthy fetuses that will come in monthly for fetal echcos starting at 20 wks.
  Interventions: Other: Maternal Hyperoxygenation
- Chonic Maternal Hyperoxygenation w/ LHH (Experimental): Mothers who have a fetus diagnosed with LHH and elect daily maternal hyperoxygenation therapy.
  Interventions: Other: Maternal Hyperoxygenation
- Acute Maternal Hyperoxygenation with LHH (Experimental): Mothers who have a fetus diagnosed with LHH and elect acute maternal hyperoxygenation challenge testing.
  Interventions: Other: Maternal Hyperoxygenation

INTERVENTIONS:
Other: Maternal Hyperoxygenation — Oxygen is given to mothers at 8L through a non-rebreather mask.
  Other Names: Oxygen
  Arms: Acute Maternal Hyperoxygenation with LHH; Chonic Maternal Hyperoxygenation w/ LHH; Healthy Fetal Controls

SUMMARY:
Heart disease is the leading cause of infant death related to birth defects. Congenital heart disease in which the left sided structures of the heart (left heart hypoplasia or LHH) are too small are among the most severe, and have some of the highest death and other complication rates.

DETAILED DESCRIPTION:
We intend to study a new, non-invasive fetal intervention to help outcomes in children with LHH. We plan to study the effect of giving oxygen to mothers who have fetuses with small left-sided structures. We specifically will evaluate if the fetal left heart valves will grow faster if the mother breathes extra oxygen on a daily basis (at least 8 hours per day). Mothers and fetuses meeting criteria will be offered to enroll in the study. All enrolled mothers will be asked to receive oxygen continuously for the rest of the pregnancy using a non-rebreather mask. At birth, we will compare the fetuses whose mothers received oxygen to historical controls. We specifically will study how fast the left heart valves have grown.

ELIGIBILITY:
Inclusion Criteria:

* Group A, C: Fetuses with hypoplastic left sided structures or at risk of coarctation of the aorta and ALL of the following

  * Any mitral annulus, aortic annulus, left ventricular end-diastolic dimension, or aortic diameter z-score less than or equal to 3.0
  * Right-left ventricular size discrepancy with no other explanation of discrepancy
  * Retrograde blood flow in the aortic arch from the ductus arteriosus
  * Left to right flow across the foramen ovale
* Group B: Healthy Fetal controls

  * Mothers undergoing screening fetal echo for family history of CHD with a normal echo.
  * Mothers undergoing fetal echocardiography for suspected heart disease with a normal echo
  * Mothers evaluated in the fetal center with normal ultrasound
* Group D:

Fetuses with hypoplastic left sided structures or at risk of coarctation of the aorta and any of the following

* Any mitral annulus, aortic annulus, left ventricular end-diastolic dimension, or aortic diameter z-score less than or equal to 2.0
* Right-left ventricular size discrepancy with no other explanation of discrepancy
* Continuous Doppler flow in the aortic arch concerning for coarctation
* Significantly less aortic flow than pulmonary artery flow
* Severe atrial septal aneurysm with possible obstruction of mitral valve flow
* Left superior vena cava to coronary sinus with dilated coronary sinus.
* Retrograde blood flow in the aortic arch from the ductus arteriosus
* Hypoplastic left heart syndrome (HLHS) and variants of HLHS
* Total anomalous pulmonary venous return

Exclusion criteria:

* Multiple gestations
* Persistent arrhythmia
* Very poor ultrasound images, defined by the inability to reliably measure/evaluate all included cardiac structures (valve annuli, branch pulmonary arteries, PFO, and arch)
* Major extra cardiac anomalies
* Aneuploidy
* Maternal conditions that may alter fetal hemodynamics, including moderate to severe HTN requiring medication in pregnancy, preeclampsia, major or unrepaired maternal congenital heart disease, obstructive sleep apnea, severe asthma (non-responsive to inhaled steroid therapy), restrictive lung disease, severe anemia, maternal chronic renal disease known placentation abnormality (complete placenta previa, accrete, or percreta), and antiphospholipid ab syndrome

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2014-01; Primary Completion 2024-04 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Aortic annular dimension | 2 years
  By fetal echo the size of the aortic annulus in mm

SECONDARY OUTCOMES:
Mitral annular dimension | years
  By fetal echo the size of the mitral valve annulus in mm

CONTACTS AND LOCATIONS:
Overall Officials: Shaine A Morris, MD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Texas Children's Hospital Pavilion for Women, Houston, Texas, United States